CLINICAL TRIAL: NCT03781648
Title: PLA Army General Hospital of Beijing
Brief Title: Water Exchange With Narrow Band Imaging on Adenoma Detection
Acronym: NBI;ADR;WE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yuqi He (Other)
Responsible Party: Sponsor-Investigator, Yuqi He, Principal Investigator, Clinical Professor, General Hospital of Beijing PLA Military Region
Organization: General Hospital of Beijing PLA Military Region (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: PLA GH-water exchange-ADR
Record Dates: First submitted 2018-12-18; First posted 2018-12-20 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Adenoma and Polyp Detection Rates
MeSH Terms: conditions — Adenoma

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WL withdrawal method (Other): Active Comparator: WL was used on withdrawal. During the insertion phase, air pump was turned off to avoid inadvertent insufflations. Water exchange with infusion pump was used to open the lumen and simultaneous suction of infused water to allow passage of the scope in clear water. Withdrawal phase done using air insufflation.
  Interventions: Diagnostic Test: NBI withdrawal method
- NBI withdrawal method (Experimental): Experimental: NBI was used on withdrawal. During the insertion phase, air pump was turned off to avoid inadvertent insufflations. Water exchange with infusion pump was used to open the lumen and simultaneous suction of infused water to allow passage of the scope in clear water. Withdrawal phase done using air insufflation.
  Interventions: Diagnostic Test: NBI withdrawal method

INTERVENTIONS:
Diagnostic Test: NBI withdrawal method — The newly available second generation of NBI using the 290 system (290-NBI) provides an at least twofold brighter image compared with the previous version
  Other Names: Water exchange

SUMMARY:
Colorectal cancer remains the third most common cause of death from cancer worldwide. The adenoma detection rate is correlated with quality of colonoscopy and risk of postcolonoscopy CRC. Low quality of bowel preparation with fecal residue and brown liquid in the colon may lower the adenoma detection rate (ADR). Optimal bowel preparation and novel approaches for colonoscopy increases the effectiveness of colonoscopic examination to improve ADR are desirable. Water exchange, which significantly increased colon cleanliness both in the right colon and the entire colon, is characterized by insertion to the cecum in clear water in lieu of gas insufflations. Water exchange led to an increase in ADR, particularly for the improvement in the right colon, providing adequate bowel preparation.

NBI is an innovative imaging technology which efficiency for the early detection of superficial cancers in the head and neck region and the esophagus had been reported previously. In the colorectal region, different results have been reported for improvement in the adenoma detection rate of NBI compared with that of WLI. All procedures were performed up to the cecum by using a high-definition colonoscope (GIF-HQ290I; Olympus Optical ) However, whether NBI in high-definition colonoscope can increase the ADR after water exchange insertion, remains to be elucidated. The aim of this study was therefore to determine whether the use of NBI system as an adjunct to water exchange insertion would improve the ADR

DETAILED DESCRIPTION:
Design: Prospective single-blinded randomized controlled trial. Patients were randomly assigned to control group or study group through a computer-based randomization list by a technician. See also inclusion and exclusion criteria.

Colonoscopy was performed using high-definition colonoscope (GIF-HQ290I) after bowel preparation. Experienced endoscopists (each with over 3000 colonoscopies performed) and fellows (performed more than 600 colonoscopies) performed all procedures. During the insertion phase, air pump was turned off to avoid inadvertent insufflations. Water exchange with infusion pump was used to open the lumen and simultaneous suction of infused water to allow passage of the scope in clear water. Suction of water can maximize cleanliness and minimize distension. Air pockets at any location of the lumen were always aspirated. In a collapsed colon, water turbulence formation at the tip of the scope facilitates residual feces removal, salvage cleansing also be provided during insertion. Simethicone was used to remove bubbles over the mucosa. Cecal intubation was defined as the passage of the scope tip beyond the ileocecal valve with visualization of the cecal appendix. After cecal intubation, as much residual water as possible was aspirated before beginning the withdrawal phase. The same endoscopist uses the same assigned method to perform tandem or back-to-back colonoscopy on all patients. After the first colonoscopic examination with the colonoscope removed from the anus, using the same entry method for insertion and the same assigned method for the second colon examination. In all arms, withdrawal lasted at least 9 minutes and was done using air insufflation to obtain adequate distension. A stopwatch was used to time the procedures, and time for polypectomy was not included.

Colon cleanliness was assessed using the Boston Bowel Preparation Scale (BBPS) and bubble scores. Cardiopulmonary function was monitored throughout, and adverse outcomes were recorded.

Study end points The primary outcome was to compare the ADR of the 290-NBI with the HD-WL. Secondary outcomes included Right and left colon Adenoma Detection Rate. Right and left colon <10 mm Adenoma Detection Rate. Mean adenomas resected per procedure. Cecal intubation rate. Cecal intubation time. Total withdrawal time. Amount of water used during the procedure. Adenoma and polyp miss rate between the two group.

ELIGIBILITY:
Inclusion Criteria:

* • Any patient ≥40 and <85 who underwent colonoscopy, does not meet exclusion criteria mentioned below and provide written informed consent will be eligible for enrolment

Exclusion Criteria:

* • (1) history of inflammatory bowel disease;(2) familial adenomatous polyposis; (3) hereditary non-polyposis colorectal cancer syndrome; (4) personal history of colorectal cancer or had previous colonic resection; (5) haemodialysis; (6) an American Society of Anaesthesiologists class III or higher; (7) antiplatelet or anticoagulant therapy 5 days before the procedure

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2018-10-20 (Actual); Primary Completion 2024-10-20 (Estimated); Study Completion 2024-10-20 (Estimated)

PRIMARY OUTCOMES:
Adenoma and polyp Detection Rate between the 290-NBI and the HD-WL group | 6 months
  Overall ADR detection rate

SECONDARY OUTCOMES:
Right and left colon Adenoma Detection Rate | 6 months
  ADR detection rate at different location
Right and left colon <10 mm Adenoma Detection Rate | 12 months
  small polyp detection rate
Mean adenomas resected per procedure | 6 months
  Total number of adenomas resected per subject
Total withdrawal time | 6 months
  Total procedure time (including time required for polyp resection or biopsy)
Amount of water used during the procedure | 6 months
  Amount of water used during insertion and withdrawal
adenoma and polyp miss rate between the two groups | 6 months
  lesion miss rate

CONTACTS AND LOCATIONS:
Overall Officials: tianyang zhang, Principal Investigator — Medical department
Locations (1):
- Department of Gastroenterology, PLA Army General Hospital, Beijing, Dongcheng District, China

IPD SHARING:
Plan to Share IPD: Undecided
After the research has been finished

REFERENCES:
- [Background] Cadoni S, Falt P, Rondonotti E, Radaelli F, Fojtik P, Gallittu P, Liggi M, Amato A, Paggi S, Smajstrla V, Urban O, Erriu M, Koo M, Leung FW. Water exchange for screening colonoscopy increases adenoma detection rate: a multicenter, double-blinded, randomized controlled trial. Endoscopy. 2017 May;49(5):456-467. doi: 10.1055/s-0043-101229. Epub 2017 Mar 10. PMID 28282689